CLINICAL TRIAL: NCT00165477
Title: Phase II Study of Lenalidomide and Radiation Therapy in Patients With Newly Diagnosed Glioblastoma Multiforme.
Brief Title: Study of Lenalidomide and XRT in Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Celgene Corporation (Industry); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); University of Virginia (Other)
Responsible Party: Patrick Wen, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-222
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Glioblastoma; Gliosarcoma; Malignant Gliomas
Keywords: Glioblastoma; Gliosarcoma; Malignant Gliomas; Radiation Therapy; IMiD; Lenalidomide
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma | interventions — Lenalidomide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lenalidomide — Given orally once a day for 21 days followed by a 1 week rest period. Subject may continue to receive study drug as long as the disease does not worsen and they experience serious side effects
  Other Names: Revlimid
Radiation: Radiation — Starting 4-7 days after the start of lenalidomide and given once a day, 5 days a week for 6-7 weeks
  Other Names: XRT

SUMMARY:
- The purpose of this study is to find out if the combination of lenalidomide and radiation therapy is effective in controlling tumor growth in patients with newly-diagnosed supratentorial glioblastoma or gliosarcoma.

DETAILED DESCRIPTION:
* Patients will receive lenalidomide orally once daily for 21 days followed by a one week rest period (this is equivalent to one cycle).
* Four to seven days from the first dose of lenalidomide, the patient will start radiation therapy for approximately 6-7 weeks.
* A neurologic exam and routine blood tests will be performed weekly while the patient is receiving radiation therapy.
* Following the 11th week of treatment a MRI/CT scan will be performed to assess the status of the tumor. If there is no change, or there is shrinkage in the size of the tumor, the treatment will continue for another 4 week cycle.
* The four week cycle will continue as long as the disease remains stable or improved and the patient does not develop intolerable side effects. A MRI/CT scan will be done every 2 cycles (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed newly-diagnosed supratentorial glioblastoma multiforme (GBM) or gliosarcoma will be eligible for this protocol.
* The patient must have recovered from the effects of surgery, post-operative infections and other complications before entry into the study.
* Diagnosis will have been established by biopsy or resection no more than 28 days prior to registration.
* If tumor resection or open biopsy was performed, cranial MRI or contrast CT must have been performed before and after surgery. Imaging within 96 h of surgery is preferred but not required.
* If needle biopsy (stereotactic) was performed, gadolinium MRI or contrast CT within 14 days prior to registration is required. A post-operative scan is not required. The use of MRI rather than CT is preferred. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement. Patients without measurable or assessable disease are eligible.
* Patients receiving steroids must be on stable or decreasing doses for at least 5 days prior to entry.
* Patients must have a plan to begin partial brain radiotherapy 4-7 days after beginning lenalidomide, and within 35 days of the surgical procedure that established the diagnosis.
* Radiotherapy must be at the Radiation Oncology Department of the registered institution.
* Patients must be willing to forego cytotoxic and non-cytotoxic drug therapy against the tumor while being treated with lenalidomide.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must be > 18 years old, and with a life expectancy > 8 weeks.
* Patients must have a Karnofsky performance status of > 60.
* Patients must have adequate bone marrow, liver, and renal function.
* Patients must be willing and able to comply with all study requirements

Exclusion Criteria:

* Patient must not have had prior cranial radiation therapy.
* Patients must not have received prior cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors. Patients who received Gliadel wafers will be excluded.
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients must not have active infection.
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have serious concurrent medical illness.
* Patient with recent thromboembolic disease (deep vein thrombosis and pulmonary embolism) are eligible if they are clinically stable and the thromboembolic event occurred more than 2 weeks prior to enrollment into this protocol.
* Patients must not have metastases below the tentorium or beyond the cranial vault.
* Patients must not have a known diagnosis of HIV, active infectious hepatitis, or chronic hepatitis.
* Patients must have no history of hypersensitivity or development of a desquamating rash while on thalidomide.
* Patients must have no prior exposure to lenalidomide.
* Previous or planned stereotactic radiosurgery or brachytherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of lenalidomide with conventional radiation therapy in the treatment of patients with newly-diagnosed supratentorial glioblastoma or gliosarcoma. | 3 years

SECONDARY OUTCOMES:
To assess the proportion of patients treated with lenalidomide and radiation therapy surviving at 12 months | 3 years
to evaluate the time to tumor progression | 3 years
the radiologic response | 3 years
to determine the safety and toxicity of the combination of lenalidomide and radiation therapy. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Virginia, Charlottesville, Virginia